CLINICAL TRIAL: NCT05631418
Title: The Children's Hospital, Zhejiang University School of Medicine, National Clinical Research Center for Child Health
Brief Title: Chinese Regional Spinal Muscular Atrophy Patient Registration Study
Status: Withdrawn | Type: Observational
Why Stopped: Due to the lack of application materials, the normal research can not be carried out for the time being.
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Shanshan Mao, Director, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: CHZhejiang
Record Dates: First submitted 2022-10-23; First posted 2022-11-30 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Recruitment
Keywords: Spinal Muscular Atrophy; long-term follow-up; quality of life; disease-modifying treatment; clinical efficacy; disease prognosis; newborn screening
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Genomic DNA may be extracted from the whole blood samples of the patients to carry out the genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objectives of this study are to obtain clinically meaningful data on the survival, outcomes, prognosis and treatment effect of all the patients with spinal muscular atrophy (SMA) 5q types 1 to 3 (according to international classification), being followed in the Children's Hospital, Zhejiang University School of Medicine since October 2019. The registry will collect retrospectively and prospectively the longitudinal data of the long-term follow-up for children patients, under real life conditions of current medical practice, in order to document the clinical evolution of patients (survival, motor, respiratory, orthopedic and nutritional and so on), the conditions of use of the treatments, the mortality rates of treated and untreated patients, the tolerance of the treatments, adverse events.

DETAILED DESCRIPTION:
The detailed objectives of this study included but not be limited to the following aspects:

1. to collect and describe overall demographic, familial, clinical, biological, and genetic characteristics of patients with 5qSMA diagnosed and treated in regions of China, by the type of SMA (type 1,2, and 3);
2. to study the impact of proactive and symptomatic medical interventions (such as bracing) and medications (disease-modifying treatment, anti-infectious, digestive, nutritional supplements, ect.) in the evolution of patients;
3. to study the long-term evolution (survival, motor and respiratory functions, spinal shape, growth and nutritional function) of 5qSMA in treated and untreated populations, by new available therapies;
4. to study the incidence and mortality rate of 5qSMA in treated and untreated populations;
5. to identify and document the different therapeutic strategies by sub-populations and by discontinuation or follow-up of treatments;
6. to evaluate prognostic factors of responses to different drug therapies;
7. to study the tolerance of treatments by type of treatments, by type of SMA and overall tolerance (including adverse events);
8. to help popularize newborn screening for SMA and pre-symptom treatment among Chinese population;
9. to get knowledge of the probable costs of care for 5qSMA patients in different groups (disease types, ages);
10. to provide needful elements to evaluate the health care costs for the disease;
11. to study the autonomy and the quality of life of patients depending on different therapies and the impact on patients' caregivers;
12. to help facilitate development of basic research on SMA in the conduct of trials on new treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Genetically confirmed 5qSMA patients through 1 to 3 types younger than 18 years old followed in our hospital since October 2019;
2. For prospective study: inform consent form signed by patient;
3. Not combined with any other genetic and metabolic diseases;

Exclusion Criteria:

1. Other type of SMA (not 5q).
2. Under guardianship or curatorship.
3. Unable to understand or cooperate with the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Genetically confirmed 5qSMA patients through 1 to 3 types younger than 18 years old followed in our hospital since October 2019 with or without disease-modifying treatment.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
World Health Organization (WHO) motor milestone change | baseline, 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  Treated and untreated patients with SMA Type 1-3: change of WHO motor milestone from baseline to 3 years to track the patients' motor functional development/status. World Health Organization motor milestone score ranges from 0 to 18. The higher the score is, the better the motor function is.
Hammersmith Infant Neurological Examination-2 (HINE-2) scale score change | baseline, 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  Treated and untreated patients with SMA Type 1-3: change of HINE-2 scale score from baseline to 3 years to help track the patients' motor functional development/status. The HINE-2 scale score ranges from 0 to 26. The higher the score is, the better the motor function is.
Self-reporting/Caregivers' reporting collection | baseline, 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  Treated and untreated patients with SMA Type 1-3: motor function change acquired from patients themselves and their caregivers. (Subjective reports were collected through interviews and no evaluation scale was used here.)
Motor function evalution-Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders(CHOP INTEND) scale | treated/untreated: baseline, 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  For children ≤ 2 years: change of CHOP INTEND scale score. The CHOP INTEND scale score ranges from 0 to 64. The higher the score is, the better the motor function is.
Motor function evalution-Hammersmith Functional Motor Scale-Expanded(HFMSE) scale | treated/untreated: baseline, 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  For children older than 2 years, ambulatory or not: Change of HFMSE scale score. The scale score ranges from 0 to 66. The higher the score is, the better the motor function is.
Motor function evalution-Revised Upper Limb Module(RULM) scale | treated/untreated: baseline, 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  For children children older than 6 years, ambulatory or not: Change of RULM (Revised Upper Limb Module) scale score. The scale score ranges from 0 to 37. The higher the score is, the better the motor function is.
Motor function evalution change-6 minutes walking test(6MWT) | treated/untreated: baseline, 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  For ambulatory individuals: added the change of 6MWT from baseline to 3 years to test exercise endurance. (The walking distance within 6 minutes is taken as the evaluation index, and there's no specific score range.)
Yearly changes of incidence and morbi-mortality-vital events | every year for 3 years
  Events of newly diagnosis, hospitalizations, recurrent infections, fractures, complications and death.
Change from baseline respiratory function | baseline(before treatment), 1 year, 2 year, 3 year
  Onset of respiratory support or change in the mode and time (including intubations).
Change from baseline digestive-nutritional function | baseline(before treatment), 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  Digestive events, onset of nutritional support or change in the mode and time and special intervention.
Change from baseline spinal scoliosis Cobb angle | baseline(before treatment), 1 year, 2 year, 3 year
  Onset of spinal deformity, or increment of over 5° in the Cobb angle (examination in supine position or in the upright position, with or without brace, with or without implant (surgery), and the change of the bone mineral density in lumbar.

SECONDARY OUTCOMES:
Pulmonary function | baseline(before treatment), 1 year, 2 year, 3 year
  Pulmonary Function Test （PFT）will be evaluated at least once per year for children > 5 years, by specifying the posture of realization of the test, lying vs sitting.
Cardiological function monitoring | baseline(before treatment), 1 year, 2 year, 3 year
  Conventional echocardiography will be evaluated to monitor the patients' cardiac function.
Body composition measurement-Lean body mass | baseline(before treatment), 1 year, 2 year, 3 year
  Lean body mass will be measured in patients older than three years by DXA or Inbody device at least once a year.
Body composition measurement-Fat mass | baseline(before treatment), 1 year, 2 year, 3 year
  Fat mass will be measured in patients older than three years by DXA or Inbody device at least once a year.
Biomarkers | baseline(before treatment), 0.5 year, 1 year, 1.5 year, 2 year, 2.5 year, 3 year
  Change of biomarkers: such as Neurofilaments.
Patients and caregivers' quality of life | baseline(before treatment), 1 year, 2 year, 3 year
  Questionary as the "PedsQL Child report/PedsQL parent report concerning child" will be used to evaluate patient's quality of life. The Pediatric Quality of Life Inventory Measurement Models (PedsQLTM) is used for this evalution. The minimum score is 0 and no specific maximum score of this scale. The higher the score is, the higher the quality of life is.

CONTACTS AND LOCATIONS:
Overall Officials: Shanshan Mao, MD, Principal Investigator — The Children's Hospital of Zhejiang University School of Medicine
Locations (1):
- The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, China